CLINICAL TRIAL: NCT04264273
Title: Intra Vitam Diagnosis of Parkinson´s Disease by Means of Submandibular Gland Needle Biopsy
Brief Title: Diagnosis of Parkinson´s Disease by Means of Submandibular Gland Needle Biopsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Principal Investigator, Joerg Spiegel, Assistant medical director, Universität des Saarlandes
Other Study IDs: 234/19
Record Dates: First submitted 2020-01-27; First posted 2020-02-11 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Parkinson Disease
Keywords: Alpha synuclein
MeSH Terms: conditions — Parkinson Disease; Parkinson Disease 4, Autosomal Dominant Lewy Body

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tissue of the submandibular gland which is obtained by means of needle biopsy from the submandibular gland
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with Parkinson´s disease.: Participants who fulfilled the diagnostic criteria of Parkinson´s disease.
- Participants without a neurological disease: 25 neurologically healthy patients of the local otolaryngological clinic, in whom submandibular gland needle biopsy was performed due to a clinical indication.

SUMMARY:
This study includes 35 PD patients who underwent submandibular gland needle biopsy. 25 neurologically healthy patients of the local otolaryngological clinic, in whom submandibular gland needle biopsy was performed due to a clinical indication, serve as controls.

DETAILED DESCRIPTION:
Parkinson´s disease (PD) is a neurodegenerative disease which is characterized by a pathological aggregation of α-synuclein. This pathological α-synuclein aggregation results in the formation of Lewy bodies which are used for the histopathological diagnosis of PD. Neuropathological post mortem studies showed that pathological aggregations of α-synuclein may occur also outside the central nervous system in PD, for example in the cardiac plexus, in the major salivary glands and the innervating cervical superior ganglion, in the minor salivary glands, in the adrenal glands and in the mesenteric and pelvic plexus. The finding of pathologically aggregated α-synuclein in the major salivary glands offers the possibility to prove PD intra vitam by means of a small transcutaneous biopsy.

A recent post mortem study in the local Department of Neuropathology found, that there was pathologically aggregated α-synuclein in 12 of 14 patients with diagnosed and neuropathologically confirmed PD, whereas there was no pathologically aggregated α-synuclein in 13 persons without PD.

The present study includes 35 PD patients who underwent submandibular gland needle biopsy. 25 neurologically healthy patients of the local otolaryngological clinic, in whom submandibular gland needle biopsy was performed due to a clinical indication, serve as controls. Immediately after the biopsy, the obtained submandibular gland tissue is transported to the local Department of Neuropathology for histopathological analysis.

ELIGIBILITY:
Inclusion Criteria: major patients with Parkinson´s disease (PD)

Exclusion Criteria:

* Missing consent to participation in the study
* Pregnancy
* Indigestibility against local anesthetic
* Increased risk of bleeding
* Therapy with an anticoagulant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unselected cohort of PD patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-02-07 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Pathologically aggregated α-synuclein in the submandibular gland. | only baseline, no further investigations.
  The biopsy was taken with a biopsy needle (diameter 14 g) which was inserted under sonographic control into one of the both submandibular glands. By means of this biopsy method, a biopsy cylinder was obtained from one submandibular gland. The biopsy cylinder which was immediately transported to the Department of Neuropathology. The whole biopsy cylinder was histopathologically investigated for pathologically aggregated alpha-synuclein. Two histopathological results are possible: presence of at least one pathologically aggregated alpha-synuclein in the obtained biopsy cylinder (positive result) or absence of any pathologically aggregated alpha-synuclein in the obtained biopsy cylinder (negative result).

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Spiegel, MD, Principal Investigator — Department of Neurology, Saarland University, D-66421 Homburg/Saar, Germany
Locations (1):
- Department of Neurology, Saarland University, Homburg/Saar, Saarland, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified individual participant data for all measures will be made available.

REFERENCES:
- [Background] Adler CH, Dugger BN, Hentz JG, Hinni ML, Lott DG, Driver-Dunckley E, Mehta S, Serrano G, Sue LI, Duffy A, Intorcia A, Filon J, Pullen J, Walker DG, Beach TG. Peripheral Synucleinopathy in Early Parkinson's Disease: Submandibular Gland Needle Biopsy Findings. Mov Disord. 2016 Feb;31(2):250-6. doi: 10.1002/mds.26476. Epub 2016 Jan 22. PMID 26799362
- [Background] Beach TG, Adler CH, Dugger BN, Serrano G, Hidalgo J, Henry-Watson J, Shill HA, Sue LI, Sabbagh MN, Akiyama H; Arizona Parkinson's Disease Consortium. Submandibular gland biopsy for the diagnosis of Parkinson disease. J Neuropathol Exp Neurol. 2013 Feb;72(2):130-6. doi: 10.1097/NEN.0b013e3182805c72. PMID 23334596
- [Background] Del Tredici K, Hawkes CH, Ghebremedhin E, Braak H. Lewy pathology in the submandibular gland of individuals with incidental Lewy body disease and sporadic Parkinson's disease. Acta Neuropathol. 2010 Jun;119(6):703-13. doi: 10.1007/s00401-010-0665-2. Epub 2010 Mar 14. PMID 20229352
- [Background] Orimo S, Uchihara T, Nakamura A, Mori F, Kakita A, Wakabayashi K, Takahashi H. Axonal alpha-synuclein aggregates herald centripetal degeneration of cardiac sympathetic nerve in Parkinson's disease. Brain. 2008 Mar;131(Pt 3):642-50. doi: 10.1093/brain/awm302. Epub 2007 Dec 13. PMID 18079166
- [Background] Spillantini MG, Schmidt ML, Lee VM, Trojanowski JQ, Jakes R, Goedert M. Alpha-synuclein in Lewy bodies. Nature. 1997 Aug 28;388(6645):839-40. doi: 10.1038/42166. No abstract available. PMID 9278044